CLINICAL TRIAL: NCT01389401
Title: Salivary Epidermal Growth Factor (EGF) Concentration Before and After Treatment of Reflux Laryngitis: Final Results
Brief Title: Salivary Epidermal Growth Factor (EGF) Concentration Before and After Treatment of Reflux Laryngitis
Status: Completed | Type: Observational
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, CLAUDIA ALESSANDRA ECKLEY, Claudia A. Eckley, MD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: cescsp179/04
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Chronic Laryngitis
Keywords: Larynx; GERD; saliva; epidermal growth factor
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngeal Diseases | interventions — Omeprazole; Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- reflux laryngitis group pre-treatment: adults with clinical suspicion of Reflux Laryngitis confirmed by 24-hour double probe esophageal monitoring who have not made use of any treatment in the past 15 days.
  Interventions: Drug: omeprazole
- study group - post treatment: adults with reflux laryngitis after 16 weeks of treatment with proton pump inhibitor (omeprazole 40 mg twice a day)and dietary/lifestyle changes that present improvement in symptoms and video laryngoscopic signs of chronic laryngitis
  Interventions: Drug: omeprazole
- control group: healthy controls paired by gender and age that do not present symptoms and videolaryngoscopic signs suggestive of reflux laryngitis
  Interventions: Drug: omeprazole

INTERVENTIONS:
Drug: omeprazole — omeprazole 40 mg twice a day for 16 weeks; dietary and lifestyle changes
  Other Names: reflux group pre-treatment; reflux group post-treatment; control group

SUMMARY:
* Saliva plays a key role in the homeostasis of the digestive tract
* The reflux of gastroesophageal contents may cause damage to the esophageal, laryngeal and pharyngeal mucosas
* There seems to be no correlation between the severity of reflux episodes and the intensity of inflammatory changes, suggesting individual protective mechanisms to refluxate exposure
* Inorganic and Organic Salivary changes have been associated to Gastroesophageal Reflux Disease (GERD) and its supraesophageal manifestations, especially reflux laryngitis (Laryngopharyngeal Reflux- LPR)
* Decreased salivary Epidermal Growth factor (EGF) concentrations have been found in patients with GERD and LPR, but it is unclear if these are primary or secondary to the disease.
* Hypothesis: The decreased salivary EGF concentrations in patients with reflux laryngitis is primary and therefore would not change after treatment and control of the disease

DETAILED DESCRIPTION:
Background & Aims: Gastroesophageal Reflux Disease (GERD) is known to affect the upper airways and may cause a variety of inflammatory changes in the pharynx and larynx. The pathophysiology of the supraesophageal forms of GERD is widely unknown. Studies have suggested decreased salivary epidermal growth factor (EGF) concentrations in patients with reflux esophagitis and laryngitis. It is however unclear if these abnormalities are primary or secondary. The aim of the current cohort study was to compare salivary EGF concentrations in adults with reflux laryngitis before and after treatment and control of the disease to that of healthy individuals. Methods: Twenty-one patients with reflux laryngitis were studied prospectively at a tertiary teaching hospital. Spontaneous whole saliva was sampled before and after a 16-week course of full dose proton pump inhibitor (PPI) twice daily and compared to that of 13 healthy controls. Salivary EGF concentrations were established using a commercially available Elisa kit.

ELIGIBILITY:
Inclusion Criteria:

* study group:

  * symptoms of reflux laryngitis (Reflux Symptom Index- RSI >13) and videolaryngoscopic signs (Reflux Finding Score - RFS >7),
  * positive 24 hour double probe esophageal PH monitoring;
* control group:

  * Reflux Symptom Index (RSI)<13
  * Reflux Finding Score (RFS) < 7

Exclusion Criteria:

* tobacco, alcohol or other inhaled drug use;
* chronic or acute rhinosinusitis;
* prior history of surgery to the digestive tract or salivary glands;
* prior or current diagnosis of head and neck or digestive tract tumors;
* chronic use of drugs known to alter salivary flow and irritate the larynx, such as, diuretics, anticonvulsants, antihistamines, and inhaled steroids

Ages: 19 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 adults with reflux laryngitis 13 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
salivary EGF concentration | 120 days
  salivary Epidermal Growth Factor (EGF) concentrations were determined with commercially available ELISA kit from whole saliva sampled before and after treatment in study group and in healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA A ECKLEY, MD, Principal Investigator — Assistant Professor Otolaryngology Department Santa Casa School of Medicine and Hospitals of São Paulo Brazil
Locations (1):
- Otolaryngology Department of Santa Casa School of Medicine and Hospitals of São Paulo Brazil, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Eckley CA, Michelsohn N, Rizzo LV, Tadokoro CE, Costa HO. Salivary epidermal growth factor concentration in adults with reflux laryngitis. Otolaryngol Head Neck Surg. 2004 Oct;131(4):401-6. doi: 10.1016/j.otohns.2004.01.020. PMID 15467608
- [Background] Sarosiek J, McCallum RW. Do salivary organic components play a protective role in health and disease of the esophageal mucosa? Digestion. 1995;56 Suppl 1:32-7. doi: 10.1159/000201299. PMID 7556968
- [Background] Rourk RM, Namiot Z, Sarosiek J, Yu Z, McCallum RW. Impairment of salivary epidermal growth factor secretory response to esophageal mechanical and chemical stimulation in patients with reflux esophagitis. Am J Gastroenterol. 1994 Feb;89(2):237-44. PMID 8304310
- [Result] Eckley CA, Rios Lda S, Rizzo LV. Salivary egf concentration in adults with reflux chronic laryngitis before and after treatment: preliminary results. Braz J Otorhinolaryngol. 2007 Mar-Apr;73(2):156-60. doi: 10.1016/s1808-8694(15)31060-0. PMID 17589721